CLINICAL TRIAL: NCT01881971
Title: Multicenter, Prospective Adaptive Response Placebo-controlled Double-blind Study Comparing Effects of Rosuvastatin Versus Placebo
Brief Title: Statins for Pulmonary and Cardiac Complications of Chronic HIV - Coordinating Center
Acronym: SPARC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alison Morris (Other)
Responsible Party: Sponsor-Investigator, Alison Morris, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO12100503; RFA-HL-12-034 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2013-04-02; First posted 2013-06-20 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: HIV Seropositivity
Keywords: HIV; lung; lipids; no lipid lowering medication; normal liver and kidney function; on stable ART regimen; not pregnant
MeSH Terms: conditions — HIV Seropositivity | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): manufactured sugar pill to mimic rouvastatin once a day for 24 weeks
  Interventions: Drug: Placebo
- Rouvastatin calcium (Experimental): Rouvastatin calcium once a day by mouth for 24 weeks.
  Interventions: Drug: Rouvastatin calcium

INTERVENTIONS:
Drug: Placebo — suger pill manufactured to mimic crestor pills
  Arms: Placebo
Drug: Rouvastatin calcium
  Other Names: Crestor
  Arms: Rouvastatin calcium

SUMMARY:
Hypothesis: Statin therapy will decrease inflammation and slow progression of cardiopulmonary abnormalities in HIV.

DETAILED DESCRIPTION:
Growing evidence indicates that chronic obstructive pulmonary disease (COPD) is an important cause of respiratory impairment in HIV+ persons and will likely increase as the HIV+ population continues to age. In the HIV-uninfected population, COPD frequently co-exists with cardiac disease including atherosclerosis and pulmonary hypertension (PH). The investigators work has demonstrated that a syndrome of "cardiopulmonary dysfunction" exists even in non-smoking or antiretroviral-treated HIV+ individuals. The investigators have found that HIV+ individuals have a high prevalence of respiratory symptoms, airflow obstruction, and diffusing capacity (DLco) abnormalities that occur concurrently with cardiac co-morbidities, including radiographic measures of atherosclerosis and elevated echocardiographic pulmonary artery pressures. This syndrome is marked by inflammation with elevated levels of cytokines and hsCRP, peripheral T-cell activation, and increased sputum neutrophils as well as elevation of NT-proBNP, a marker of heart strain. Importantly, the investigators have shown that DLco impairment and elevated NT-proBNP are significant independent predictors of mortality in HIV, indicating that cardiopulmonary dysfunction is likely highly clinically relevant and identifies a vulnerable population in whom the investigators lack effective interventions.

Statins have anti-inflammatory effects in the lung and vasculature that might benefit cardiopulmonary dysfunction in HIV. These agents have a long history of clinical use in cardiovascular disease and are currently being investigated as disease-modifying drugs for HIV, COPD, and PH. In preliminary analyses, the investigators have found that HIV+ individuals who received statin therapy within the past year were significantly less likely to have impaired DLco and had lower pulmonary artery pressures, lower NT-proBNP, lower peripheral cytokines, and fewer sputum neutrophils despite being older and having a greater smoking history than those not using statins.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented in medical record at any time prior to study entry.
* Men and women age18 years to 80 years.
* Presence of COPD (FEV1/FVC<0.70 or DLco≤80% predicted)
* No lipid-lowering medication (prescription or non-prescription) within 60 days prior to study entry. This includes all statin drugs, omega-3-fatty acids/fish oil (if dose > 1 g/day), red yeast rice (any dose), and niacin products (e.g., niacin, nicotinic acid, vitamin B3; if dose of >100 mg/day)
* Normal liver and kidney function test at screening visit:
* Liver function: ALT 7 to 55 U/L; AST 8 to 48 U/L; ALP 45 to 115 U/L; Bilirubin 0.1 to 1.0 mg/dL; GGT 9 to 48 U/L; LDH 122 to 222 umol/L; PT 8.3 to 10.8 seconds
* Kidney function: BUN 8-20 mg/dl. Creatinine 0.8-1.2 mg/dl for males and 0.6-0.9 mg/dl for females. GFR normal results range from 90 - 120 mL/min/1.73 m2.) Participants will be on a stable ART regimen (i.e. no change in agents) with either suppressed HIV viral level or <50 viral level for at least 3 months.
* If smoker, not planning on quitting smoking during the study period. If non-smoker, not planning on starting smoking during the study period.
* Able to provide informed consent.
* Able to participate in study procedures based on the investigator's assessment.
* For women of reproductive potential, negative urine pregnancy test and willingness to use birth control during study period (see Contraception requirements).
* Ability and willingness to complete all tests.
* Participant in MACS, Women's Interagency Health Study, or Attendee of UPMC HIV / AIDS Program.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Known allergy/sensitivity or any hypersensitivity to HMG CoA reductase inhibitors, prior history of myopathy, rhabdomyolysis, or intolerance of statin therapy.
* Currently receiving a statin or should be taking a statin based on clinical criteria.
* Concurrent use of Coumadin.
* History of liver disease.
* Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
* Diagnosis of asthma with normal diffusing capacity.
* History of diabetes mellitus requiring medication of hemoglobin A1C>6.5% on screening laboratories.
* Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
* Hospitalization within 4 weeks prior to study entry.
* Use of antibiotics within 4 weeks of study entry.
* Uncontrolled hypertension at screening visit (systolic > 160 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
* Active cancer requiring systemic chemotherapy or radiation.
* Active infection of lungs, brain, or abdomen.
* Use of anti-inflammatory agents (such as aspirin), immunomodulators (e.g., interleukins, interferons, cyclosporine) or immunosuppressive medications within 60 days prior to study entry. Routine vaccinations are allowed if administered at least 7 days prior to study entry.
* Use of azole antifungals, erythromycin, or amiodarone.
* More than weekly use of magnesium hydroxide.
* The intention to quit smoking during the study period.
* Alcoholism defined as >35 drinks per week or that will impair ability to complete study investigations in the opinion of the investigator.
* Active (within the past 6 months) intravenous drug use or that will impair ability to complete study investigations in the opinion of the investigator.
* Use of other investigational agents within 90 days of study entry or planning on entering another therapy trial during study period.
* No use of inhaled corticosteroids (beta-agonists are allowed).
* Viral load above 50 in past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in inflammatory markers - hsCRP | 24 weeks
  To assess change in hsCRP after 24 weeks of therapy with rosuvastatin

SECONDARY OUTCOMES:
effect of rosuvastatin on pulmonary and cardiac status by use of cIMT/FMD/ Vascular studies are a measure of preclinical atherosclerosis and predicts future cardiovascular events and mortality | 2 years
  noninvsive Vascular cIMT, FMD and Glycocalyx will be measured at the beginning and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Morris, MD, MS, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of California, Los Angelos, Los Angeles, California
  - University of California, SF, San Francisco, California
  - University of Pittsburgh department of medicine division of Pulmonary, Allergy and Critical Care medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Morris A, Fitzpatrick M, Bertolet M, Qin S, Kingsley L, Leo N, Kessinger C, Michael H, Mcmahon D, Weinman R, Stone S, Leader JK, Kleerup E, Huang L, Wisniewski SR. Use of rosuvastatin in HIV-associated chronic obstructive pulmonary disease. AIDS. 2017 Feb 20;31(4):539-544. doi: 10.1097/QAD.0000000000001365. PMID 27941393